CLINICAL TRIAL: NCT04695535
Title: Chemotherapy With Anlotinib in Advanced Cervical Cancer: A Prospective, Single-arm Study
Brief Title: Chemotherapy With Anlotinib in Advanced Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yang Shen (Other)
Responsible Party: Sponsor-Investigator, Yang Shen, Deputy Director of Zhongda Hospital, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: ZhongdaH-YShen
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Anlotinib; Chemotherapy; Advanced Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy with Anlotinib: Patients received chemotherapy with Anlotinib.

SUMMARY:
STUDY HYPOTHESIS: The primary hypothesis is whether chemotherapy with Anlotinib improves overall survival in advanced cervical cancer.

TRIAL DESIGN: The study is a prospective, single-arm, observational clinical study. The study will be performed on an intent-to-treat population. All the enrolled patients received chemotherapy with Anlotinib.

PRIMARY ENDPOINT: Overall survival, defined as the observed length of life from entry into the study to death from any cause or the date of last contact.

DETAILED DESCRIPTION:
Patients with advanced (metastatic, persistent, and recurrent) cervical cancer will be recruited from Zhongda Hospital. Only patients who treated with paclitaxel plus nedaplatin will be included in the analysis. All patients receive paclitaxel (135-175mg /m^2) and nedaplatin (100 mg/m^2) infusion on day 1, and then take Anlotinib 12mg/d orally on day 7-21, every 3 weeks. Once patients reached CR or PR, Anlotinib was continued on 12mg/d maintenance therapy until disease progression or unacceptable toxicity was noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced (metastatic, persistent, and recurrent) cervical cancer confirmed by imaging and unsuitable for surgery and radiotherapy .
* Eastern Cooperative Oncology Group (ECOG) Performance Score(PS) 0-1
* Estimated life expectancy > 3 months
* Adequate bone marrow function: hemoglobin > 90 g/L, absolute neutrophil count(ANC) > 1.5 × 10^9/L, platelet > 80 × 10^9/L);
* Adequate hepatic function: total bilirubin < 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<2.5×ULN or <5×ULN for patients with liver metastases;
* Adequate renal function: serum creatinine < 1.5 × ULN or creatinine clearance rate (CCR) >60 mL/min;
* Adequate cardiac function: left ventricular ejection fraction (LVEF) > 50%.

Exclusion Criteria:

* Preexisting thyroid disease, thyroid function cannot be maintained in the normal range after treatment;
* Have used other anti-VEGF or VEGFR-targeted drugs or received immunotherapy;
* A history of major surgical treatment within 4 weeks, radiotherapy within 3 weeks, and concurrent chemoradiotherapy within 6 weeks;
* Receiving hormone or immunosuppressive therapy for various reasons;
* Inability to swallow oral medication;
* Any malabsorption;
* Diseases diagnosed as severe or uncontrollable within 6 months prior to the first day of treatment.
* Participate in clinical trials of other antitumor drugs within 28 days prior to the start of study treatment;
* The patient has comorbidities that may endanger the patient's safety or affect the patient's ability to complete the study.
* According to the researcher's judgment, the patient has an accompanying disease that may jeopardize the patient's safety or affect the patient's ability to complete the study in the investigator's judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced (metastatic, persistent, and recurrent) cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years
  The time from the first day of treatment until death from any cause

SECONDARY OUTCOMES:
Progression-free survival | Up to 3 years
  The time from the first day of treatment until disease progression or death from any cause, or as the date of the last follow-up.
Incidence of Adverse Events [Safety and Tolerability] | Up to 3 years
  Adverse Events were assessed according to the National Cancer Institute's Common Toxicity Criteria (CTCAE) version 4.0.
The average score of FACT-Cx TOI [Functional Assessment] | Up to 3 years
  The HRQL instruments used in this trial were the Functional Assessment of Cancer Therapy-Cervix (FACT-Cx) Trial Outcome Index (TOI), for which a higher score indicates better HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No